CLINICAL TRIAL: NCT00004313
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Dehydroepiandrosterone Replacement for Primary Adrenal Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11822; UCSD-1062
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Addison's Disease
Keywords: Addison's disease; endocrine disorders; rare disease; primary adrenal insufficiency
MeSH Terms: conditions — Addison Disease; Endocrine System Diseases; Rare Diseases | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: dehydroepiandrosterone

SUMMARY:
OBJECTIVES:

I. Determine the efficacy of dehydroepiandrosterone (DHEA), an androgen replacement hormone, for patients with primary adrenal insufficiency (Addison's disease).

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by age.

Patients are randomly assigned to androgen replacement therapy with daily dehydroepiandrosterone (DHEA) or placebo for 6 months. All patients may receive 6 additional months of DHEA following randomized therapy.

Women on hormonal replacement therapy may receive concurrent conjugated estrogens or oral medroxyprogesterone.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Primary adrenal insufficiency (Addison's disease) Serum dehydroepiandrosterone less than 0.5 nmol/L --Prior/Concurrent Therapy-- No concurrent investigational drug Stable glucocorticoid/mineralocorticoid dose over past year required --Patient Characteristics-- Hepatic: No hepatic disease Cardiovascular: No vascular disease No thrombotic disorder No angina No elevated blood pressure on 2 readings taken 15 minutes apart in 1 visit, i.e.: Systolic greater than 165 mm Hg OR Diastolic greater than 95 mm Hg Other: No clinically significant medical abnormality No gallbladder disease No malignancy No estrogen- or androgen-dependent neoplasia Benign prostatic hyperplasia eligible No other endocrine disease Controlled thyroid disease with normal thyroid-stimulating hormone eligible Mammogram required within 1 year prior to entry for women aged 40 and over No clinically significant abnormality No undiagnosed vaginal or uterine bleeding within 6 months prior to entry Pap smear required within 1 year prior to entry No dysplasia (squamous intraepithelial lesion low-grade or higher)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1995-08

CONTACTS AND LOCATIONS:
Overall Officials: Samuel S. C. Yen, Study Chair — University of California, Los Angeles